CLINICAL TRIAL: NCT04088370
Title: Peripheral Blood Mononuclear Cells Response In Healthy Controls, Heavy Drinkers, and Patients With Alcoholic Hepatitis
Status: Recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Srinivasan Dasarathy, Staff Physician, The Cleveland Clinic
Other Study IDs: 19-1041
Record Dates: First submitted 2019-09-11; First posted 2019-09-12 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Alcoholic Hepatitis
MeSH Terms: conditions — Hepatitis, Alcoholic | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral Blood Mononuclear Cells, ethylenediaminetetraacetic acid (EDTA) plasma and serum will be collected
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Alcoholic Hepatitis: No intervention-blood draw only
  Interventions: Other: Blood Draw
- Healthy Controls: No intervention- blood draw only
  Interventions: Other: Blood Draw
- Healthy Heavy Drinkers: No intervention- blood draw only
  Interventions: Other: Blood Draw

INTERVENTIONS:
Other: Blood Draw — Blood Draw Only

SUMMARY:
Inflammatory responses in response to alcohol have been identified as contributing to the development of alcoholic hepatitis. The inflammatory response including that to LippoPolySaccharide is known to lead to progression of alcoholic liver disease. In addition to the inflammatory response mitochondrial perturbations exist and redox homeostasis is altered in patients with alcoholic hepatitis. Though this is known there have been very few studies targeting mitochondrial function in Peripheral Blood Mononuclear Cells (PBMCs). We plan to collect 50 milliliters of blood from healthy control patients so that we can compare the data to that of patients with alcoholic hepatitis and those who are heavy drinkers without liver disease. In addition to studying mitochondrial function we will investigate cytokine response, as well as fatty acid metabolism, glucose, and insulin measurements

ELIGIBILITY:
Inclusion of Subjects with Alcoholic Hepatitis (AH):

*diagnosis of AH either by imaging, biochemical values or liver biopsy as well as drinking history

Inclusion Heavy Drinking Controls:

*heavy alcohol drinking will be defined as >40 g/day or >280g/week on average for women and >60 g/day or >420 g/week on average for men for a minimum of 6 months [6] and within the 4 weeks prior to study enrollment.

Exclusion Criteria for all groups

* inability or unwillingness to sign informed consent
* cancer
* autoimmune disease that in the opinion of the PI will confound study data

Control subjects (drinking and non drinking) must meet the following criteria:

* INR < 1.4
* total bilirubin levels must <3
* no prior history of known alcoholic liver disease
* absence of hepatosplenomegaly (from physical examination or radiographic imaging) or stigmata of liver disease.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with alcoholic hepatitis as diagnosed by liver biopsy, imaging, or biochemical values with noted encounter in Cleveland Clinic Electronic Medical Record,
  Heavy Drinking Controls - patients who lack any evidence (biochemical, imaging, and/or biopsy) of alcoholic liver disease who consume >40 g/day or >280g/week on average for women and >60 g/day or >420 g/week on average for men for a minimum of 6 months
  Healthy Controls - patients without any form of liver disease nd do not meet the criteria for "Heavy Drinking Controls"
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-10-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Quantify mitochondrial respiration | 1 day
  Mitochondrial Respiration will be quantified by using a standard substrate, uncoupler, inhibitor titration protocol using high resolution respirometry

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States